CLINICAL TRIAL: NCT07092826
Title: Obsessive-Compulsive Disorder: Formal and Content Modalities, Factors Involved in Loss of Insight, Role of Trauma, and Correlations With Schizophrenia Spectrum Disorders
Brief Title: Obsessive-Compulsive Disorder: Insight, Trauma, and Links to Schizophrenia Spectrum Disorders
Status: Active, not recruiting | Type: Observational
Sponsor: Matteo Tonna (Other)
Collaborators: San Raffaele University Hospital, Italy (Other)
Responsible Party: Sponsor-Investigator, Matteo Tonna, Associate Professor of Psychiatry, University of Parma, Azienda Ospedaliero-Universitaria di Parma
Organization: Azienda Ospedaliero-Universitaria di Parma (Other)
Other Study IDs: UNIPR-OCD-INSIGHT-290525-V1
Record Dates: First submitted 2025-06-03; First posted 2025-07-30 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Obsessive-Compulsive Disorder (OCD); Schizophrenia and Schizophrenia Spectrum Psychosis
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Schizophrenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Psychopathological assessment and non-invasive multisensory stimulation — This intervention consists of a non-invasive, cross-sectional assessment involving standardized psychopathological interviews and multisensory stimulation tasks (auditory, tactile, and combined). It is designed to explore formal and content-related features of obsessive-compulsive symptoms, insight levels, and trauma-related correlates in patients with OCD and schizophrenia spectrum disorders. No pharmacological treatment or experimental therapy is administered as part of this study.

SUMMARY:
This study aims to better understand Obsessive-Compulsive Disorder (OCD) by examining the types and patterns of OCD symptom presentation. The investigators seek to determine how these symptoms impact overall daily functioning.

The study will also explore factors contributing to loss of insight in individuals with OCD, focusing on the potential roles of trauma, personality traits, and disorder severity. This may assist in identifying subgroups of patients who respond more favorably to treatment.

Additionally, the study will investigate how individuals with OCD and schizophrenia spectrum symptoms respond to combined sensory stimuli (e.g., auditory and tactile). The goal is to determine whether these responses are associated with specific brain processing patterns, trauma history, or characteristics of compulsive behavior. Insights from this research may help clarify why certain individuals develop repetitive behaviors such as checking and rituals.

Participants will be adults aged 18 to 65 diagnosed with OCD or schizophrenia spectrum disorders. Recruitment will occur through psychiatric clinics in Parma. Participation requires signed informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Obsessive-Compulsive Disorder (OCD) and/or Schizophrenia Spectrum Disorder according to DSM-5 criteria (APA, 2013), as determined by a structured clinical interview (SCID-5-CV) (First et al., 2016).
* Age between 18 and 65 years.
* Participant agreement to take part in the study (informed consent).

Exclusion Criteria:

* General medical condition that may be related to the psychiatric disorder.
* Alcohol or substance dependence or abuse.
* Cognitive impairment (score below 25 on the Mini Mental State Examination).

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The patients are affiliated with the facilities of the Integrated Department of Mental Health and Pathological Addictions (DAI-SMDP) of the Parma Local Health Authority (AUSL Parma)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Yellbrown (Y-BOCS) Score | Baseline (single evaluation session)
  Assessment of obsessive-compulsive symptom severity using the Yellow-Brown Obsessive-Compulsive Scale (Y-BOCS). The total score ranges from 0 to 40, with higher scores indicating more severe symptoms. This scale is a clinician-administered questionnaire evaluating obsessions and compulsions

SECONDARY OUTCOMES:
Childhood Trauma Questionnaire-Short Form (CTQ-SF) Total Score | Baseline (single evaluation session)
  Measurement of childhood trauma exposure using the Childhood Trauma Questionnaire-Short Form (CTQ-SF), a self-report questionnaire with scores ranging from 25 to 125. Higher scores indicate greater levels of reported childhood trauma
Simultaneity Judgement Task (SJ) Performance | Approximately 15 minutes during the pre-training session
  Assessment of audio-tactile simultaneity perception using paired auditory and tactile stimuli presented with varying temporal delays. Participants are asked to judge whether the stimuli occur simultaneously. The task includes multiple trials with systematically varied stimulus onset asynchronies. Performance is defined as the proportion of correct simultaneity judgments, reflecting multisensory temporal integration abilities
Simultaneity Judgement Training (SJT) Performance | Approximately 30-45 minutes during the training session
  Evaluation of training-induced improvements in multisensory temporal integration through a task where participants receive real-time feedback on their simultaneity judgments. A staircase procedure adjusts the delay between stimuli based on participant responses. Performance is measured as improvement in simultaneity judgment accuracy and reduced temporal thresholds from pre- to post-training sessions

OTHER OUTCOMES:
Structural Analysis of Rituals | Baseline (single evaluation session)
  Behavioral analysis of ritual videos conducted with ethnographic software, which breaks down rituals into elementary behavioral units classified into three categories: functional, non-functional, and displaced. The measure quantifies the frequency of each behavioral unit category to assess the complexity and structure of rituals. Frequency counts of behavioral units per category (functional, non-functional, displaced). Baseline and follow-up video recordings.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - University of Parma, Parma, Emilia-Romagna
  - Università degli Studi di Parma - Dipartimento di Medicina e Chirurgia, Parma

REFERENCES:
- [Background] Insel TR, Akiskal HS. Obsessive-compulsive disorder with psychotic features: a phenomenologic analysis. Am J Psychiatry. 1986 Dec;143(12):1527-33. doi: 10.1176/ajp.143.12.1527. PMID 3789205
- [Background] Innamorati M, Erbuto D, Venturini P, Fagioli F, Ricci F, Lester D, Amore M, Girardi P, Pompili M. Factorial validity of the Childhood Trauma Questionnaire in Italian psychiatric patients. Psychiatry Res. 2016 Nov 30;245:297-302. doi: 10.1016/j.psychres.2016.08.044. Epub 2016 Aug 16. PMID 27567192
- [Background] Huber G, Gross G. The concept of basic symptoms in schizophrenic and schizoaffective psychoses. Recenti Prog Med. 1989 Dec;80(12):646-52. PMID 2697899
- [Background] Henderson JG Jr, Pollard CA. Three types of obsessive compulsive disorder in a community sample. J Clin Psychol. 1988 Sep;44(5):747-52. doi: 10.1002/1097-4679(198809)44:53.0.co;2-2. PMID 3263989
- [Background] Hemmings SM, Lochner C, van der Merwe L, Cath DC, Seedat S, Stein DJ. BDNF Val66Met modifies the risk of childhood trauma on obsessive-compulsive disorder. J Psychiatr Res. 2013 Dec;47(12):1857-63. doi: 10.1016/j.jpsychires.2013.08.012. Epub 2013 Sep 2. PMID 24050777
- [Background] Heins M, Simons C, Lataster T, Pfeifer S, Versmissen D, Lardinois M, Marcelis M, Delespaul P, Krabbendam L, van Os J, Myin-Germeys I. Childhood trauma and psychosis: a case-control and case-sibling comparison across different levels of genetic liability, psychopathology, and type of trauma. Am J Psychiatry. 2011 Dec;168(12):1286-94. doi: 10.1176/appi.ajp.2011.10101531. Epub 2011 Sep 28. PMID 21955935
- [Background] Hagen K, Solem S, Opstad HB, Hansen B, Hagen R. The role of metacognition and obsessive-compulsive symptoms in psychosis: an analogue study. BMC Psychiatry. 2017 Jun 29;17(1):233. doi: 10.1186/s12888-017-1392-1. PMID 28662637
- [Background] Gothelf D, Aharonovsky O, Horesh N, Carty T, Apter A. Life events and personality factors in children and adolescents with obsessive-compulsive disorder and other anxiety disorders. Compr Psychiatry. 2004 May-Jun;45(3):192-8. doi: 10.1016/j.comppsych.2004.02.010. PMID 15124149
- [Background] Goodman WK, Price LH, Rasmussen SA, Mazure C, Delgado P, Heninger GR, Charney DS. The Yale-Brown Obsessive Compulsive Scale. II. Validity. Arch Gen Psychiatry. 1989 Nov;46(11):1012-6. doi: 10.1001/archpsyc.1989.01810110054008. PMID 2510699
- [Background] Goodman WK, Price LH, Rasmussen SA, Mazure C, Fleischmann RL, Hill CL, Heninger GR, Charney DS. The Yale-Brown Obsessive Compulsive Scale. I. Development, use, and reliability. Arch Gen Psychiatry. 1989 Nov;46(11):1006-11. doi: 10.1001/archpsyc.1989.01810110048007. PMID 2684084
- [Background] Goldman HH, Skodol AE, Lave TR. Revising axis V for DSM-IV: a review of measures of social functioning. Am J Psychiatry. 1992 Sep;149(9):1148-56. doi: 10.1176/ajp.149.9.1148. PMID 1386964
- [Background] Garcia-Perez MA, Alcala-Quintana R. Response errors explain the failure of independent-channels models of perception of temporal order. Front Psychol. 2012 Apr 4;3:94. doi: 10.3389/fpsyg.2012.00094. eCollection 2012. PMID 22493586
- [Background] Fujisaki W, Nishida S. Audio-tactile superiority over visuo-tactile and audio-visual combinations in the temporal resolution of synchrony perception. Exp Brain Res. 2009 Sep;198(2-3):245-59. doi: 10.1007/s00221-009-1870-x. Epub 2009 Jun 5. PMID 19499212
- [Background] Fontenelle JM, Harrison BJ, Santana L, Conceicao do Rosario M, Versiani M, Fontenelle LF. Correlates of insight into different symptom dimensions in obsessive-compulsive disorder. Ann Clin Psychiatry. 2013 Feb;25(1):11-6. PMID 23376865
- [Background] Fontenelle IS, Fontenelle LF, Borges MC, Prazeres AM, Range BP, Mendlowicz MV, Versiani M. Quality of life and symptom dimensions of patients with obsessive-compulsive disorder. Psychiatry Res. 2010 Sep 30;179(2):198-203. doi: 10.1016/j.psychres.2009.04.005. Epub 2010 May 18. PMID 20483484
- [Background] Foa EB, Kozak MJ, Goodman WK, Hollander E, Jenike MA, Rasmussen SA. DSM-IV field trial: obsessive-compulsive disorder. Am J Psychiatry. 1995 Jan;152(1):90-6. doi: 10.1176/ajp.152.1.90. PMID 7802127
- [Background] Ettelt S, Grabe HJ, Ruhrmann S, Buhtz F, Hochrein A, Kraft S, Pukrop R, Klosterkotter J, Falkai P, Maier W, John U, Freyberger HJ, Wagner M. Harm avoidance in subjects with obsessive-compulsive disorder and their families. J Affect Disord. 2008 Apr;107(1-3):265-9. doi: 10.1016/j.jad.2007.08.017. Epub 2007 Sep 12. PMID 17854908
- [Background] Erzegovesi S, Cavallini MC, Cavedini P, Diaferia G, Locatelli M, Bellodi L. Clinical predictors of drug response in obsessive-compulsive disorder. J Clin Psychopharmacol. 2001 Oct;21(5):488-92. doi: 10.1097/00004714-200110000-00006. PMID 11593074
- [Background] Endicott J, Spitzer RL, Fleiss JL, Cohen J. The global assessment scale. A procedure for measuring overall severity of psychiatric disturbance. Arch Gen Psychiatry. 1976 Jun;33(6):766-71. doi: 10.1001/archpsyc.1976.01770060086012. PMID 938196
- [Background] Eisen JL, Mancebo MA, Pinto A, Coles ME, Pagano ME, Stout R, Rasmussen SA. Impact of obsessive-compulsive disorder on quality of life. Compr Psychiatry. 2006 Jul-Aug;47(4):270-5. doi: 10.1016/j.comppsych.2005.11.006. Epub 2006 Apr 19. PMID 16769301
- [Background] Eisen JL, Phillips KA, Coles ME, Rasmussen SA. Insight in obsessive compulsive disorder and body dysmorphic disorder. Compr Psychiatry. 2004 Jan-Feb;45(1):10-5. doi: 10.1016/j.comppsych.2003.09.010. PMID 14671731
- [Background] Eisen JL, Rasmussen SA, Phillips KA, Price LH, Davidson J, Lydiard RB, Ninan P, Piggott T. Insight and treatment outcome in obsessive-compulsive disorder. Compr Psychiatry. 2001 Nov-Dec;42(6):494-7. doi: 10.1053/comp.2001.27898. PMID 11704942
- [Background] Eisen JL, Rasmussen SA. Obsessive compulsive disorder with psychotic features. J Clin Psychiatry. 1993 Oct;54(10):373-9. PMID 8262879
- [Background] Eilam D. From an animal model to human patients: An example of a translational study on obsessive compulsive disorder (OCD). Neurosci Biobehav Rev. 2017 May;76(Pt A):67-76. doi: 10.1016/j.neubiorev.2016.12.034. PMID 28434589
- [Background] Dettore D, Pozza A, Coradeschi D. Does time-intensive ERP attenuate the negative impact of comorbid personality disorders on the outcome of treatment-resistant OCD? J Behav Ther Exp Psychiatry. 2013 Dec;44(4):411-7. doi: 10.1016/j.jbtep.2013.04.002. Epub 2013 May 15. PMID 23770674
- [Background] de Silva P, Marks M. The role of traumatic experiences in the genesis of obsessive-compulsive disorder. Behav Res Ther. 1999 Oct;37(10):941-51. doi: 10.1016/S0005-7967(98)00185-5. PMID 10472711
- [Background] De Berardis D, Campanella D, Gambi F, Sepede G, Salini G, Carano A, La Rovere R, Pelusi L, Penna L, Cicconetti A, Cotellessa C, Salerno RM, Ferro FM. Insight and alexithymia in adult outpatients with obsessive-compulsive disorder. Eur Arch Psychiatry Clin Neurosci. 2005 Oct;255(5):350-8. doi: 10.1007/s00406-005-0573-y. Epub 2005 Feb 21. PMID 15711867
- [Background] Cromer KR, Schmidt NB, Murphy DL. An investigation of traumatic life events and obsessive-compulsive disorder. Behav Res Ther. 2007 Jul;45(7):1683-91. doi: 10.1016/j.brat.2006.08.018. Epub 2006 Oct 25. PMID 17067548
- [Background] Conroy E, Degenhardt L, Mattick RP, Nelson EC. Child maltreatment as a risk factor for opioid dependence: Comparison of family characteristics and type and severity of child maltreatment with a matched control group. Child Abuse Negl. 2009 Jun;33(6):343-52. doi: 10.1016/j.chiabu.2008.09.009. Epub 2009 May 23. PMID 19477004
- [Background] Cheng YF, Chen VC, Yang YH, Chen KJ, Lee YC, Lu ML. Risk of schizophrenia among people with obsessive-compulsive disorder: A nationwide population-based cohort study. Schizophr Res. 2019 Jul;209:58-63. doi: 10.1016/j.schres.2019.05.024. Epub 2019 May 24. PMID 31133461
- [Background] Cederlof M, Lichtenstein P, Larsson H, Boman M, Ruck C, Landen M, Mataix-Cols D. Obsessive-Compulsive Disorder, Psychosis, and Bipolarity: A Longitudinal Cohort and Multigenerational Family Study. Schizophr Bull. 2015 Sep;41(5):1076-83. doi: 10.1093/schbul/sbu169. Epub 2014 Dec 15. PMID 25512596
- [Background] Catapano F, Perris F, Fabrazzo M, Cioffi V, Giacco D, De Santis V, Maj M. Obsessive-compulsive disorder with poor insight: a three-year prospective study. Prog Neuropsychopharmacol Biol Psychiatry. 2010 Mar 17;34(2):323-30. doi: 10.1016/j.pnpbp.2009.12.007. Epub 2009 Dec 16. PMID 20015461
- [Background] Catapano F, Sperandeo R, Perris F, Lanzaro M, Maj M. Insight and resistance in patients with obsessive-compulsive disorder. Psychopathology. 2001 Mar-Apr;34(2):62-8. doi: 10.1159/000049282. PMID 11244376
- [Background] Bulli F, Melli G, Cavalletti V, Stopani E, Carraresi C. Comorbid Personality Disorders in Obsessive-Compulsive Disorder and Its Symptom Dimensions. Psychiatr Q. 2016 Jun;87(2):365-76. doi: 10.1007/s11126-015-9393-z. PMID 26442944
- [Background] Briggs ES, Price IR. The relationship between adverse childhood experience and obsessive-compulsive symptoms and beliefs: the role of anxiety, depression, and experiential avoidance. J Anxiety Disord. 2009 Dec;23(8):1037-46. doi: 10.1016/j.janxdis.2009.07.004. Epub 2009 Jul 8. PMID 19635653
- [Background] Boyer P, Lienard P. Why ritualized behavior? Precaution Systems and action parsing in developmental, pathological and cultural rituals. Behav Brain Sci. 2006 Dec;29(6):595-613; discussion 613-50. doi: 10.1017/s0140525x06009332. PMID 17918647
- [Background] Black DW, Noyes R Jr, Pfohl B, Goldstein RB, Blum N. Personality disorder in obsessive-compulsive volunteers, well comparison subjects, and their first-degree relatives. Am J Psychiatry. 1993 Aug;150(8):1226-32. doi: 10.1176/ajp.150.8.1226. PMID 8328568
- [Background] Bernstein DP, Ahluvalia T, Pogge D, Handelsman L. Validity of the Childhood Trauma Questionnaire in an adolescent psychiatric population. J Am Acad Child Adolesc Psychiatry. 1997 Mar;36(3):340-8. doi: 10.1097/00004583-199703000-00012. PMID 9055514
- [Background] Bey K, Lennertz L, Riesel A, Klawohn J, Kaufmann C, Heinzel S, Grutzmann R, Kathmann N, Wagner M. Harm avoidance and childhood adversities in patients with obsessive-compulsive disorder and their unaffected first-degree relatives. Acta Psychiatr Scand. 2017 Apr;135(4):328-338. doi: 10.1111/acps.12707. Epub 2017 Feb 3. PMID 28160276
- [Background] Baer L, Jenike MA. Personality disorders in obsessive compulsive disorder. Psychiatr Clin North Am. 1992 Dec;15(4):803-12. PMID 1461797
- [Background] Alonso P, Lopez-Sola C, Real E, Segalas C, Menchon JM. Animal models of obsessive-compulsive disorder: utility and limitations. Neuropsychiatr Dis Treat. 2015 Aug 4;11:1939-55. doi: 10.2147/NDT.S62785. eCollection 2015. PMID 26346234
- [Background] Alonso P, Menchon JM, Segalas C, Jaurrieta N, Jimenez-Murcia S, Cardoner N, Labad J, Real E, Pertusa A, Vallejo J. Clinical implications of insight assessment in obsessive-compulsive disorder. Compr Psychiatry. 2008 May-Jun;49(3):305-12. doi: 10.1016/j.comppsych.2007.09.005. Epub 2007 Dec 21. PMID 18396191
- [Background] Afifi TO, Mather A, Boman J, Fleisher W, Enns MW, Macmillan H, Sareen J. Childhood adversity and personality disorders: results from a nationally representative population-based study. J Psychiatr Res. 2011 Jun;45(6):814-22. doi: 10.1016/j.jpsychires.2010.11.008. Epub 2010 Dec 10. PMID 21146190
- [Background] Adam Y, Meinlschmidt G, Gloster AT, Lieb R. Obsessive-compulsive disorder in the community: 12-month prevalence, comorbidity and impairment. Soc Psychiatry Psychiatr Epidemiol. 2012 Mar;47(3):339-49. doi: 10.1007/s00127-010-0337-5. Epub 2011 Feb 2. PMID 21287144

DOCUMENTS (3):
  • Study Protocol (2025-05-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT07092826/Prot_003.pdf
  • Informed Consent Form: Informative Document (2025-05-17): https://cdn.clinicaltrials.gov/large-docs/26/NCT07092826/ICF_001.pdf
  • Informed Consent Form: Informed Consent Form (2023-01-28): https://cdn.clinicaltrials.gov/large-docs/26/NCT07092826/ICF_002.pdf